CLINICAL TRIAL: NCT03315078
Title: Lentiviral Gene Transfer for Treatment of Children Older Than 2 Years of Age With X-Linked Severe Combined Immunodeficiency
Acronym: LVXSCID-OC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-I-0007
Record Dates: First submitted 2017-10-16; First posted 2017-10-19 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: X-Linked Combined Immunodeficiency Diseases
MeSH Terms: conditions — X-Linked Combined Immunodeficiency Diseases | interventions — Fibroblast Growth Factor 7; Busulfan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Gene-Modified CD34+ HSCs (Experimental): Participants will receive palifermin on Days -6, -5, and -4 and then busulfan on Days -3 and -2. On Day 0, participants will undergo the gene transfer treatment with infusion of the gene-modified CD34+ HSCs. They will receive palifermin on Days 1, 2, and 3.
  Interventions: Biological: CD34+ HSCs transduced with the lentivirus vector, VSV-G pseudotyped CL20-4i-EF1α-hγc-OPT; Drug: Palifermin; Drug: Busulfan

INTERVENTIONS:
Biological: CD34+ HSCs transduced with the lentivirus vector, VSV-G pseudotyped CL20-4i-EF1α-hγc-OPT — Administered by intravenous (IV) infusion
Drug: Palifermin — Administered by IV infusion at a dose of 60 mg/kg/day
Drug: Busulfan — Administered by IV infusion at a dose of approximately 3 mg/kg per day

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of lentiviral gene transfer treatment at restoring immune function to participants with X-linked severe combined immunodeficiency (XSCID) who are 2 to 40 years of age, and have significant impairment of immunity.

DETAILED DESCRIPTION:
This study will evaluate the safety and effectiveness of lentiviral gene transfer treatment at restoring immune function to participants with X-linked severe combined immunodeficiency (XSCID) who are 2 to 40 years of age, and have significant impairment of immunity. XSCID is a severe genetic condition of the immune system.

Participants in this study will be treated at the National Institutes of Health (NIH) Clinical Center.

Before the gene transfer treatment, a participant's own CD34+ hematopoietic stem cells (HSCs) will have been or will be collected from the participant's blood or bone marrow. When the participant has the required number of HSCs harvested, then the participant's HSCs will be grown in tissue culture and exposed to the lentiviral gene transfer vector containing the corrective gene (VSV-G pseudotyped CL20-4i-EF1α-hγc-OPT). These gene corrected HSCs will be administered by intravenous (IV) infusion to the participant. To increase engraftment of the corrected HSCs, participants will receive a chemotherapy drug called busulfan on 2 days before the gene transfer treatment. Participants will also receive palifermin, which helps prevent mucositis, which is the main side effect from the busulfan.

After the gene transfer treatment, participants will be monitored to see if the treatment is safe and whether their immune system improves. Participants will be followed at frequent intervals for the first 2 years, and less frequently thereafter so that the effectiveness in restoration of immune function and the safety of the treatment can be evaluated. Additional safety follow-up may occur through Year 15.

ELIGIBILITY:
Inclusion Criteria:

* A proven mutation in the common gamma chain gene as defined by direct sequencing of patient DNA
* Human leukocyte antigen (HLA) typing of the patient will have been performed before enrollment
* No available HLA matched sibling donor as determined before enrollment.
* Must be between 2 and 40 years of age and weigh 10 kg
* If previously transplanted, must be 18 months post-hematopoietic stem cell transplant (HSCT)
* Expected survival of at least 120 days.
* Documented to be negative for HIV infection by genome polymerase chain reaction (PCR)
* The patient must be judged by the primary evaluating physician to have a suitable family and social situation consistent with ability to comply with protocol procedures and the long-term follow-up requirements.
* Medical lab data (historical) of severe B cell dysfunction (low or absent immunoglobulin G [IgG] levels, failed immune response to vaccines); OR demonstrated requirement for intravenous gamma globulin (IVIG) (significant drop over 3 to 6 weeks between peak and trough IgG levels).
* Must be willing to have blood and tissue samples stored. IN ADDITION, patients must satisfy the following Laboratory Criteria AND Clinical Criteria:
* Laboratory Criteria: (at least 1 must be present)

  * CD4+ lymphocytes: absolute number less than or equal to 50% of the lower limit of normal (LLN)
  * CD4+CD45RA+ lymphocytes: absolute number less than or equal to 50% of the LLN OR T-cell receptor excision circles (TRECs) less than or equal to 5% of normal for age.
  * Memory B Cells: absolute number less than or equal to 50% of LLN
  * Serum immunoglobulin M (IgM) less than normal for age
  * Natural killer (NK) cells: absolute number less than or equal to 50% of LLN
  * Lymphocyte proliferative response to each of 2 mitogens, phytohemagglutinin (PHA) and concanavalin A (ConA), is less than or equal to 25% compared with a normal control.
  * Molecular spectratype analysis- absent or very oligoclonal (1-3 dominant peaks) in greater than or equal to 6 of the 24 Vbeta T-cell receptor families.
* Clinical Criteria: (at least 1 must be present)
* i. Infections (not including molluscum, warts or mucocutaneous candidiasis; see vii and viii below): 3 significant new or chronic active infections during the 2 years preceding evaluation for enrollment, with each infection accounting for one criteria. Infections are defined as an objective sign of infection (fever greater than 38.3^0C [101^0F] or neutrophilia or pain/redness/swelling or radiologic/ultrasound imaging evidence or typical lesion or histology or new severe diarrhea or cough with sputum production). In addition to one or more of these signs/symptoms of possible infection, there also must be at least 1 of the following criteria as evidence of the attending physician's "intent to treat" a significant infection (a. and b.) or objective evidence for a specific pathogen causing the infection (c.)

  * a. Treatment (not prophylaxis) with systemic antibacterial, antifungal or antiviral antibiotics 14 days OR
  * b. Hospitalization of any duration for infection OR
  * c. Isolation of a bacteria, fungus, or virus from biopsy, skin lesion, blood, nasal washing, bronchoscopy, cerebrospinal fluid or stool likely to be an etiologic agent of infection
* ii. Chronic pulmonary disease as defined by:

  * a. Bronchiectasis by x-ray computerized tomography OR
  * b. Pulmonary function test (PFT) evidence for restrictive or obstructive disease that is 60% of Predicted for Age OR
  * c. Pulse oximetry 94% in room air (if patient is too young to comply with performance of pulmonary function tests [PFTs]).
* iii. Gastrointestinal enteropathy:

  * a. Diarrhea-watery stools 3 times per day (of at least 3 months duration that is not a result of infection as defined in criterion number i. above) OR
  * b. Endoscopic evidence (gross and histologic) for enteropathy (endoscopy will only be performed if medically indicated) OR
  * c. Other evidence of enteropathy or bacterial overgrowth syndrome: including malabsorption of fat soluble vitamin(s), abnormal D-xylose absorption, abnormal hydrogen breath test, evidence of protein losing enteropathy (for example increasingly high or frequent dosing of intravenous gamma globulin supplement required to maintain blood IgG level).
* iv. Poor nutrition: Requires gastrostomy tube (G-tube) or intravenous feeding supplement to maintain weight or nutrition.
* v. Auto- or allo-immunity: Examples must include objective physical findings that include, but are not limited to any one of alopecia, severe rashes, uveitis, joint pain with redness or swelling or limitation of movement that is not a result of infection, lupus-like lesions, and granulomas (Does not include auto- or allo-immune enteropathy which is criterion iii). Where possible and appropriate, diagnosis will be supported by histopathology or other diagnostic modality.
* vi. Failure to grow in height: 3rd percentile for age
* vii. Skin molluscum contagiosum OR warts (this criterion is satisfied if molluscum consists of 10 lesions or there are two or more lesions at each of two or more widely separated anatomic sites; or there are 3 warts at different anatomic sites at the same time; or the patient has both molluscum and warts)
* viii. Mucocutaneous candidiasis (chronic oral thrush or candida esophagitis or candida intertriginous infection or candida nail infections; must be culture positive to satisfy this criterion)
* ix. Hypogammaglobulinemia: requires regular IgG supplementation

Exclusion Criteria:

* Any current or pre-existing hematologic malignancy
* Current treatment with any chemotherapeutic agent (becomes eligible if not on treatment for at least 3 months)
* Documented HIV-1 infection
* Documented active Hepatitis B infection
* Childhood malignancy (occurring before 18 years of age) in the patient or a first degree relative, or previously diagnosed known genotype of the subject conferring a predisposition to cancer (no DNA or other testing for cancer predisposition genes will be performed as part of the screen for this protocol)

Ages: 2 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 13 (Estimated)
Dates: Start 2012-04 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Level of autologous transduced T-lymphocytes with functional γc | Measured through Year 2
  Defined by their appearance and expansion in peripheral blood
Incidence of serious side effects due to lentiviral gene transfer | Measured through Year 15
  As determined by whether participants experience any grade 3 or greater toxicity that is directly attributed to the gene therapy procedure
Distribution of integration sites of the lentiviral vector in reconstituted peripheral blood cells | Measured through Year 15
  Based on statistical analysis

CONTACTS AND LOCATIONS:
Overall Officials: Suk See DeRavin, M.D., Ph.D, Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- Laboratory of Host Defenses (LHD), National Institute of Allergy and Infectious Diseases (NIAID), National Institutes of Health (NIH), Bethesda, Maryland, United States